CLINICAL TRIAL: NCT06171789
Title: A Phase 1/2 Study of PRO1107 in Patients With Advanced Solid Tumors
Brief Title: PRO1107 in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Genmab has decided to discontinue the clinical development of GEN1107 as the overall benefit-risk profile no longer supports continuation
Sponsor: Genmab (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCT1107-01; CTR20242075 (Other: Chinadrugtrials); PRO1107-01 (Other: Secondary Protocol ID)
Record Dates: First submitted 2023-11-29; First posted 2023-12-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Cancer; Ovarian Cancer; Triple Negative Breast Cancer; GastroEsophageal Cancer; Non-small Cell Lung Cancer; Urothelial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Transitional Cell

STUDY DESIGN:
Intervention Model Description: Modified toxicity probability interval (mTPI)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GEN1107 (Experimental): GEN1107 monotherapy in escalating doses in Part A and at the dose level in Part B.
  Interventions: Drug: GEN1107

INTERVENTIONS:
Drug: GEN1107 — IV infusion of GEN1107

SUMMARY:
This is a global, open-label, multicenter Phase 1/2 study to evaluate the safety, tolerability, pharmacokinetics (PK), and antitumor activity of GEN1107 (PRO1107) in participants with advanced solid tumors. This study consists of 2 parts, Part A: dose escalation and dose level expansion, and Part B: tumor specific expansion.

DETAILED DESCRIPTION:
This is a Phase 1/2 study of GEN1107, a protein tyrosine K 7 (PTK7) targeted antibody-drug conjugate (ADC), to evaluate the safety, tolerability, PK, and antitumor activity of GEN1107 in participants with advanced solid tumors, including ovarian cancer, endometrial cancer, triple negative breast cancer, non-small cell lung cancer, gastroesophageal cancer, and urothelial cancer. This study consists of 2 parts, Part A: Dose Escalation and Dose Level Expansion and Part B: Tumor Specific Expansion.

In Part A, GEN1107 will be administered in different dosing regimens via intravenous (IV) infusion.

Part B will be initiated at a dose level based on a comprehensive analysis of safety, tolerability, clinical PK, pharmacodynamics (PD) and activity data from Part A in up to 4 different tumor-specific cohorts of up to 40 participants per cohort.

Participants will continue to receive study treatment until the first instance of disease progression, unacceptable toxicity, investigator decision, consent withdrawal, study termination by the Sponsor, pregnancy, or death.

ELIGIBILITY:
Inclusion Criteria

Part A:

* Pathologically confirmed diagnosis of one of the following tumor types:
* Ovarian cancer (epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer)
* Endometrial cancer (any subtype excluding sarcoma)
* Triple negative breast cancer (TNBC)
* Non-small cell lung cancer (NSCLC)

  * Metastatic or unresectable locally advanced, recurrent, disease not amenable to further local therapy following prior systemic therapies known to confer clinical benefit.

Part B:

* Participants must have a histologically or cytologically confirmed metastatic or unresectable solid malignancy as specified below:

  * Ovarian cancer
  * TNBC
  * Endometrial cancer
  * NSCLC
* Measurable disease at baseline as defined per RECIST, Version 1.1

Exclusion Criteria

* Prior treatment with anti-PTK7-directed therapy.
* Had progressive disease as best response while on treatment with an auristatin (eg, a vedotin or pelidotin)- based ADC as the most recent line of therapy.
* History of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Exceptions are malignancies with a negligible risk of metastasis or death (eg, 5-year overall survival [OS] ≥90%)
* Known active central nervous system metastases, including carcinomatous meningitis. Participants with brain metastases may participate provided the metastases have been treated and are stable for at least 4 weeks prior to the first dose of study drug, they have no new or enlarging brain metastases and have discontinued corticosteroids prescribed for symptoms associated with brain metastases for at least 7 days prior to the first dose of study drug. Participants with a history of brain metastases, suspected new brain metastases, or a diagnosis of NSCLC or breast cancer should have a computed tomography (CT)/ magnetic resonance imaging (MRI) scan of the brain at screening.
* Participants with active or chronic corneal disorders, history of corneal transplantation, or any clinically significant corneal disease that prevents adequate monitoring of potential drug-induced keratopathy. Note: Participants with other active ocular conditions requiring ongoing therapy and/or monitoring must be discussed with the sponsor prior to enrollment.

Additional protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Through end of treatment, up to approximately 1 year
  Type, incidence, severity, seriousness, and relatedness of adverse events.
Number of Participants with Dose Limiting Toxicities (DLTs) | Day 1 up to a maximum of Day 28
  Incidence of dose limiting toxicities.

SECONDARY OUTCOMES:
Objective Response Rate | Through end of treatment, up to approximately 1 year
  Participants who achieve partial or complete response per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria.
Disease Control Rate | Through end of treatment, up to approximately 1 year
  Participants who achieve stable disease, partial or complete response per RECIST v1.1 criteria.
Progression-free Survival | Up to approximately 18 months
  Time from start of treatment to first documented disease progression or death.
Duration of Objective Response | From date of enrollment until the date of first documented disease progression or date of study withdrawal, whichever came first, assessed up to 12 months
  Time from the first documentation of an objective tumor response (complete response or partial response) to the first documented tumor progression or death.
Pharmacokinetic Parameter Area Under the Curve (AUC) for GEN1107 | Varying timepoints through end of treatment, up to approximately 1 year
  Measure of GEN1107 AUC in plasma.
Pharmacokinetic Parameter Maximum Concentration (Cmax) for GEN1107 | Varying timepoints through end of treatment, up to approximately 1 year
  Measure of the Cmax of GEN1107 in plasma.
Pharmacokinetic Parameter Time to Maximum Concentration (Tmax) for GEN1107 | Varying timepoints through end of treatment, up to approximately 1 year
  Measure of the Tmax of GEN1107 in plasma.
Pharmacokinetic Parameter Apparent Terminal Half-life (t1/2) for GEN1107 | Varying timepoints through end of treatment, up to approximately 1 year
  Measure of t1/2 of GEN1107 in plasma.
Pharmacokinetic Parameter Trough Concentration (Ctrough) for GEN1107 | Varying timepoints through end of treatment, up to approximately 1 year
  Measure of the Ctrough of GEN1107 in plasma.
Number of Participants with Anti-drug Antibodies (ADAs) | Varying timepoints through end of treatment, up to approximately 1 year
Cancer Antigen 125 (CA-125) Response per Gynecological Cancer Intergroup (GCIG) Criteria for Ovarian Cancer | Varying timepoints through end of treatment, up to approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Genmab
Locations (7):
- United States (6):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Florida Cancer Specialists, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - SCRI Oncology Partners, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - START Mountain Cancer Center, Salt Lake City, Utah
- Institution of Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No